CLINICAL TRIAL: NCT07020182
Title: Efficacy Of Inpatient Pulmonary Rehabilitation Program In Elderly Patients With Acute Exacerbation Of COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Marwa Mohammed, Lecturer of physical therapy,Beni-suef University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INPATIENT COPD REHABILITATION
Record Dates: First submitted 2025-05-10; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: COPD Received PR; Elderly (People Aged 65 or More); COPD; COPD Acute Exacerbation
Keywords: Elderly patients with acute exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A prospective supervised RCT (Randomized Controlled Trial) will be done include elderly COPD patients assigned randomly into two groups; Group A performed physical therapy program, and Group B is control group completed two daily sessions from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The codes were determined by using serially numbered block size will be kept in sealed and opaque envelopes in a locked office
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A will perform physical therapy program (Experimental): Study group In this study we will study the impact of exercise training include breathing exercise, low-load resistance exercise (15%-30% of 1 repetition maximum (1-RM) as tolerated), aerobic training in the form of walking exercise under supervision of physiotherapist.In patients exercise tolerance, dyspnea, fatigue, and time to discharge from hospital.
  The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  Interventions: Other: physical therapy program
- Group B will the control group (No Intervention): control group

INTERVENTIONS:
Other: physical therapy program — Group A will performed a physical therapy program that completed two daily sessions till discharge from the hospital .Exercise training starts from randomisation until hospital discharge,and administered twice per day, seven times per week. The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  Arms: Group A will perform physical therapy program

SUMMARY:
The study aimed to identify the effect of early pulmonary rehabilitation in elderly patients with Acute exacerbation (AE) of COPD (AECOPD) in exercise tolerance, dyspnea, sleep quality, fatigue, and time to discharge from hospital.

DETAILED DESCRIPTION:
A prospective supervised RCT (Randomized Controlled Trial) will be done include elderly COPD patients assigned randomly into two groups; Group A performed Physical therapy program, and Group B is control group completed two daily sessions from day 1 of hospital admission till discharge from the hospital .The study duration will be 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute exacerbation of COPD in both gender
* Patient older than 65 years
* Patient with clear consciousness
* Patients had been diagnosed with shortness of breath or dyspnea that was not caused by heart disease, pneumothorax, or pulmonary edema

Exclusion Criteria:

* Patient with systolic blood pressure lower than 90 mmHg
* Patient with an unstable psychological status, hemoptysis, pneumothorax, pulmonary edema

Ages: 65 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  The 6 minute walk test(6MWT)in meter to asses exercise tolerance

SECONDARY OUTCOMES:
Dyspnea | The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  (The Modified Medical Research Council (mMRC )scale to assess Dyspnea)
Length of hospital stay(LOS) | The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  (Number of days to assess length of stay in hospital (LOS) from admission to hospital to discharge from hospital)
Fatigue level | The study will be start from day 1 of hospital admission till discharge from the hospital.The study duration will be 12 weeks
  Fatigue Severity Scale (FSS)to assess fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed, phd, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of Medicine for Girls- Al-Azhar-University, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT07020182/Prot_ICF_000.pdf